CLINICAL TRIAL: NCT01787994
Title: A Phase I, Open Label, Dual Cohort, Single Center Study to Evaluate the Safety, Tolerability and Immunogenicity of Autologous CD4 T Cells Modified With a Retroviral Vector Expressing the MazF Endoribonuclease Gene in Patients With HIV
Brief Title: Redirected MazF-CD4 Autologous T Cells for HIV Gene Therapy
Acronym: MazF
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 815441
Record Dates: First submitted 2013-01-31; First posted 2013-02-11 (Estimated); Last update posted 2019-08-30 (Actual); Status verified 2019-08

CONDITIONS: HIV

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Experimental): Cohort 1: HIV-1-positive women and men ≥18 years with a CD4 count > 350 cells/mm3, HIV-1-RNA levels undetectable by ultrasensitive HIV PCR Abbott assay. Subjects with HIV-1 RNA < 400 copies/mL are also eligible; however, the HIV-1 RNA must be < 50 copies/mL within 60 days prior to study entry based on the Abbott assay. Subjects with intermittent isolated episodes of detectable low level viremia (> 50 but <1,000 copies RNA/mL; blips) will be eligible.
  There should be at least 2 documented HIV-1 RNA assays, one drawn >3 months before study entry, one drawn <3 months before study entry. Subjects should be on HAART (no changes to treatment within 4 weeks of study entry) for at least 3 months.
  Cohort 1 subjects will receive a single dose of MazF-T cells.
  Interventions: Genetic: Autologous CD4+ T cells genetically modified with a retroviral vector expressing the MazF endoribonuclease gene (MazF-T), given via intravenous infusion.
- Cohort 2 (Experimental): Cohort 2: HIV-1-positive men and women ≥18 years with a CD4 count > 450 cells/mm3, having well controlled HIV replication on HAART. The subjects should have a CD4 nadir ≥200 cells/mm3. Subjects in Cohort 2 will participate in a 16 week analytical treatment interruption beginning 2 weeks after T cell infusion.
  Cohort 2 subjects will receive a single dose of MazF-T cells.
  Interventions: Genetic: Autologous CD4+ T cells genetically modified with a retroviral vector expressing the MazF endoribonuclease gene (MazF-T), given via intravenous infusion.

INTERVENTIONS:
Genetic: Autologous CD4+ T cells genetically modified with a retroviral vector expressing the MazF endoribonuclease gene (MazF-T), given via intravenous infusion.

SUMMARY:
This is an open label, dual cohort study evaluating safety, tolerability and immunogenicity of redirected CD4+ T cells in HIV subjects.

ELIGIBILITY:
Inclusion Criteria:

1. HIV-1 infection, as documented by a rapid HIV test or any FDA-approved HIV-1 enzyme or chemiluminescence immunoassay (E/CIA) test kit and confirmed by Western blot at any time prior to study entry. Alternatively, if a rapid HIV test or any FDA-approved HIV-1 enzyme or chemiluminescence immunoassay (E/CIA) test kit is not available, two HIV-1 RNA values >2000 copies/mL at least 24 hours apart performed by any laboratory that has CLIA certification, or its equivalent, may be used to document infection.
2. Antiretroviral medication

   * Cohort 1: Subjects on HAART (no changes to treatment within 4 weeks of study entry) for at least 3 months.
   * Subjects on HAART (no changes to treatment within 4 weeks of study entry) for at least 3 months.
3. Plasma HIV viremia

   * Cohort 1: HIV-1-positive men and women >18 years of age with HIV-1-RNA levels undetectable by ultrasensitive HIV PCR Abbott assay at screening. Also eligible are subjects with HIV-1 RNA < 400 copies/mL; however, the HIV-1 RNA must be < 50 copies/mL within 60 days prior to study entry based on the Abbott assay. Subjects with intermittent isolated episodes of detectable low level viremia (> 50 but <1,000 copies RNA/mL; blips) will be eligible. There should be at least 2 documented HIV-1 RNA assays, one drawn >3 months before study entry, one drawn <3 months before study entry.
   * Cohort 2: HIV-1-positive men and women >18 years of age with HIV-1-RNA levels undetectable by ultrasensitive HIV PCR assay at screening. Note: Due to sensitivity issues using the Roche Assay and the fact that we cannot control the HIV testing technique prior to enrollment, we decided to consider subjects with HIV-1 RNA < 400 copies/mL; however, the HIV-1 RNA must be undetectable within 60 days prior to study entry based on the ultrasensitive HIV PCR assay. Subjects with intermittent isolated episodes of detectable low level viremia (> 50 but <1,000 copies RNA/mL; blips) will be eligible. There should be at least 2 documented HIV-1 RNA assays: one drawn >3 months before study entry, one drawn <3 months before study entry.
4. CD4 counts

   * Cohort 1: Subjects with CD4 counts >350 cells/mm3.
   * Cohort 2: Subjects with CD4 counts of at least 450 cells/mm3 at screening. Note: CD4 nadir in Cohort 2 must be above 200 cells/mm3.
5. Adequate venous access and no other contraindications for leukapheresis.
6. Laboratory values obtained within 60 days prior to entry.

   * Hemoglobin: ≥ 10.0 (males); ≥ 9.5 (females) g/dL
   * Absolute neutrophil count (ANC): ≥ 1000/mm3
   * Platelet count: ≥ 75,000/mm3
   * Serum creatinine: ≤ 1.5 mg/dL (133μ mol/L)
   * Aspartate aminotransferase (AST) or alanine aminotransferase (ALT): ≤ 2.5 times the upper limit of normal (ULN).
7. Subjects must be willing to comply with study-mandated evaluations. Rectal biopsy procedures are optional.
8. Be male or female, 18 years of age and older.
9. Ability and willingness of subject to provide informed consent.
10. Have a Karnofsky Performance Score of 70 or higher.

Exclusion Criteria:

1. No history of opportunistic infections or neoplasm.
2. Concomitant acute or chronic hepatitis B (surface antigen positive) or hepatitis C infection. If HCV antibody test is positive, an HCV RNA test will be performed. If both HCV tests (antibody and RNA) are positive, the subjects will be excluded from study. If HCV antibody test is positive, but HCV RNA test is negative, subject can enroll. Results should be obtained no more than 30 days prior to screening.
3. History of cancer or malignancy, with the exception of successfully treated basal cell or squamous cell carcinoma of the skin.
4. 4.2.4 History or any features on physical examination indicative of active or unstable cardiac disease or hemodynamic instability.
5. History or any features on physical examination indicative of a bleeding diathesis.
6. Have been previously treated with any HIV experimental vaccine within 6 months prior to screening, or any previous gene therapy using an integrating vector.
7. Use of chronic corticosteroids, hydroxyurea, or immunomodulating agents (e.g., interleukin-2, interferon-alpha or -gamma, granulocyte colony stimulating factors, etc.) within 30 days prior to study entry.
8. Breast-feeding, pregnant, or unwilling to use acceptable methods of birth control.
9. Use of aspirin, dipyrdamole, warfarin or any other medication that is likely to affect platelet function or other aspects of blood coagulation during the 2-week period prior to leukapheresis.
10. Active drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements.
11. Serious illness requiring systemic treatment and/or hospitalization within 30 days prior to study entry.
12. Asymptomatic abnormal baseline serum chemistry elevations. Note: Asymptomatic baseline serum chemistry elevations in total or indirect bilirubin in subjects receiving atazanavir or indinavir is not exclusionary. Asymptomatic baseline serum chemistry elevations in LFTs, lipase and creatinine due to HAART medication are not exclusionary, when in the opinion of the investigator, the abnormalities are not attributable to intrinsic hepatorenal disease. Such elevations must be due to HAART.
13. Receipt of a vaccination within 30 days prior to study entry.
14. Have an allergy or hypersensitivity to study product excipients (human serum albumin, DMSO and Dextran 40).
15. For Cohort 2: CD4 nadir below 200 cells/mm3.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-12 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
The number of subjects with adverse events following a single dose of MazF transduced cells. Safety will be assessed by reviewing adverse events at 24 hours, 72 hours and 7, 14, 21 days, 4 weeks and 2, 3 and 6 months post infusion. | 3 years
Feasibility will be assessed by counting the number of manufacturing failures. | Day 0

SECONDARY OUTCOMES:
Antiviral effects will be monitored in veremic subjects of Cohort 2. The anti-viral effect of infusion will be determined by comparing the viral loads pre-infusion and post-infusion | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Infectious Diseases & HIV Medicine at Drexel University College of Medicine, Philadelphia, Pennsylvania, United States